CLINICAL TRIAL: NCT03914313
Title: Effects of Robotic Neurorehabilitation Plus Virtual Reality on Attention Process and Executive Functions in Patients With Chronic Stroke: a Randomized Controlled Trial
Brief Title: Robotics Plus VR in Improving Cognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Principal Investigator, Rocco Salvatore Calabrò, Professor, IRCCS Centro Neurolesi Bonino Pulejo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13/19
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Cognition Disorders
Keywords: Lokomat; Robotic rehab; Executive function; VR
MeSH Terms: conditions — Cognition Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Robotic Treatment plus VR (Experimental): The patients included will be divided into three groups of 30 patients each. In this group patients will undergo a rehabilitation training with the Lokomat Pro, in which the exoskeleton device is equipped with a VR screen. The rehabilitation protocol consists of 24 training sessions (3 sessions per week, for 8 weeks, each session lasting about 45 minutes). Lokomat will be used to improve gait, whereas motor and cognitive function will be normally trained by using conventional neurorehabilitation. Patients will be evaluated at baseline (T0), immediately (T1) and after 3.month (T2) of treatment.
  Interventions: Device: Robotic Treatment plus VR
- Robotic treatment without VR (Active Comparator): The patients included will be divided into three groups of 30 patients each. In this group patients will undergo a rehabilitation training with the Lokomat-Nanos, in which the exoskeleton device is equipped with a screen with a visual feedback (but not virtual reality). The rehabilitation protocol consists of 24 training sessions (3 sessions per week, for 8 weeks, each session lasting about 45 minutes). The Lokomat-Nanos will be used to improve gait, whereas motor and cognitive function will be normally trained by using conventional neurorehabilitation. Patients will be evaluated at baseline (T0), immediately (T1) and after 3.month (T2) of treatement.
  Interventions: Device: Robotic Treatment plus VR
- Conventional treatment (Active Comparator): The patients included will be divided into three groups of 30 patients each. In this group patients will undergo a conventional gait rehabilitation. The rehabilitation protocol consists of 24 training sessions (3 sessions per week, for 8 weeks, each session lasting about 45 minutes). Beside conventional overground training for gait, motor and cognitive function will be normally trained by using conventional neurorehabilitation. Patients will be evaluated at baseline (T0), immediately (T1) and after 3.month (T2) of treatement.
  Interventions: Device: Robotic Treatment plus VR

INTERVENTIONS:
Device: Robotic Treatment plus VR — The patients included will be divided into three groups of 30 patients each. In this group patients will undergo a rehabilitation training with the Lokomat-Pro, in which the exoskeleton device is equipped with a screen with virtual reality. The rehabilitation protocol consists of 24 training sessions (3 sessions per week, for 8 weeks, each session lasting about 45 minutes). The Lokomat-Pro will be used to improve gait, whereas motor and cognitive function will be normally trained by using conventional neurorehabilitation. Patients will be evaluated at baseline (T0), immediately (T1) and after 3.month (T2) of treatment.

SUMMARY:
Stroke can be classified as ischemic, i.e. due to the lack of blood flow, and haemorrhagic, caused by bleeding. Stroke results in focal signs and symptoms, with a devastating impact on a patient and his family. Although robotic rehabilitation is very useful in improving motor function, there is no a clear evidence on its role in improving cognitive abilities, which are often compromised in stroke patients.

To this end, the investigators designed a randomized controlled experimental study on stroke patients, with the aim of evaluating the effects of robotic neurorehabilitation using Lokomat with and without virtual reality on cognitive functioning in stroke patients, compared to traditional therapy.

ELIGIBILITY:
Inclusion Criteria:

Neurological diagnosis of stroke in the post-acute phase (3 months from the acute event); age between 40 and 80; and Caucasian ethnicity; a FIM motor score equal to or greater than 30 and moderate to mild cognitive impairment (MoCA> 18); Fugl-Meyer scale score of> 18;

Exclusion Criteria:

Patients with a history of concomitant neurodegenerative diseases or brain surgery; severe cognitive or language impairment; systemic, bone or joint disorders; presence of disabling sensory alterations; concomitant medical and psychiatric illness that could interfere with VR training.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2019-11-10 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Frontal Assessment Battery | 3 months
  This is a tool is used to examine global frontal abilities

SECONDARY OUTCOMES:
Trial Making Test | 3 months
  This is a tool is used to measure the attention process, and attentive shifting.

CONTACTS AND LOCATIONS:
Overall Officials: Rocco S Calabrò, Study Chair — IRCCS Centro Neurolesi
Locations (1):
- IRCCS Centro Neurolesi "Bonino-Pulejo", Messina, Italy

IPD SHARING:
Plan to Share IPD: Undecided